CLINICAL TRIAL: NCT02482116
Title: Malaria and Pneumonia in Children Under the Age of Five Years Old Presenting to Primary Healthcare Centres in Benin City, Nigeria: a Comparison of Early Diagnostic Approaches
Brief Title: A Comparison of Diagnostic Approaches for Malaria and Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Collaborators: University of Benin (Other)
Responsible Party: Sponsor
Other Study IDs: HA.577/Vol. II/126
Record Dates: First submitted 2015-06-22; First posted 2015-06-26 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Malaria; Pneumonia
Keywords: malaria; pneumonia; Nigeria; IMCI; diagnosis
MeSH Terms: conditions — Malaria; Pneumonia; Disease | interventions — Guidelines as Topic; X-Rays; Rapid Diagnostic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: malaria or pneumonia diagnosis — Diagnostic approaches for malaria (lay diagnosis, as per IMCI guidelines by trained primary healthcare workers, clinical diagnosis by medically qualified doctor, rapid diagnostic tests, Giemsa microscopy); Diagnostic approaches for pneumonia (lay diagnosis, as per IMCI guidelines by trained primary healthcare workers, clinical diagnosis by medically qualified doctor, chest x-ray)
  Other Names: Integrated Management of Childhood Illness (IMCI) guidelines; Giemsa microscopy; Chest x-ray; Rapid diagnostic test for malaria; Lay-diagnosis of malaria & pneumonia

SUMMARY:
This research investigates the diagnostic accuracy of various diagnostic approaches for malaria and pneumonia in under-five children presenting to primary healthcare centres in Benin City, Nigeria.

DETAILED DESCRIPTION:
Of the preventable and treatable diseases, both malaria and pneumonia are significant contributors to under-five mortality in Nigeria. To reduce the burden of these diseases, the Integrated Management of Childhood Illness (IMCI) guidelines were developed by the World Health Organisation (WHO) to be used at first point of contact (e.g., primary healthcare centres) with children under the age of five years old. Preliminary literature review suggests that although interventions based on numerous diagnostic approaches have been trialed, burden from malaria and pneumonia remains unacceptably high in Nigeria, suggesting limited effectiveness of existing approaches. Therefore, this study aims to compare the accuracy of different early diagnostic approaches used in the community(for e.g. the WHO Integrated Management of Childhood Illness (IMCI) guidelines versus the gold standard diagnostic tests comprising microscopy in malaria and chest radiography in pneumonia) in children under the age of five years presenting with suspected malaria and pneumonia to primary healthcare centres in Benin City, Edo State of Nigeria.

The research will compare the accuracy of these various diagnostic approaches using measures such as sensitivity, specificity, positive predictive value, negative predictive value, and area under the receiver operating characteristic curve. The research will also assess patient outcomes like complications, hospitalisation and death following a diagnosis of either pneumonia or malaria in all study participants as well as costs associated with malaria and pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Suspected malaria (symptoms reported by caregiver that are consistent with malaria: high temperature, chills and no other probable diagnosis)
* Suspected pneumonia (fever, cough, shortness of breath/difficulty in breathing, with or without chills and no other probable diagnosis)
* Willingness of caregiver to provide written or verbal consent in the presence of a witness.

Exclusion Criteria:

None

Ages: 2 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population are children aged 2 months to four years old who are residents in the catchment local government area of study primary healthcare centres in Benin City, Edo State, Nigeria.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2015-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Malaria confirmed by microscopy (yes/no) | Participants will be assessed within an average period of 24 hours of presenting to study primary healthcare centres
  This is the gold standard diagnosis for malaria and will be used to assess the accuracy of other diagnostic approaches
Pneumonia confirmed by chest x-ray (yes/no) | Participants will be assessed within an average period of 48 hours of presenting to study primary healthcare centres
  This is the gold standard test for pneumonia and will be used to assess the accuracy of other diagnostic approaches

SECONDARY OUTCOMES:
Hospitalisation (yes/no) | Within 30 days of first consultation
  This will be assessed for all study participants with either a malaria or pneumonia diagnosis as part of an epidemiological study
Death (yes/no) | Within 30 days of first consultation
  This will be assessed for all study participants with either a malaria or pneumonia diagnosis as part of an epidemiological study

CONTACTS AND LOCATIONS:
Overall Officials: Kelly O Elimian, MSc, Principal Investigator — University of Nottingham & University of Benin; Puja R Myles, PhD, Study Director — University of Nottingham; Catherine Pritchard, PhD, Study Director — University of Nottingham; Ayebo Sadoh, PhD, Study Director — University of Benin
Locations (1):
- Health Services Department, University of Benin, Benin City, Edo, Nigeria